CLINICAL TRIAL: NCT07152691
Title: Establishing a Computational Model for a Non-Invasive Swallowing Monitoring Device: A Pilot Study
Brief Title: Non-Invasive Swallowing Monitoring Device
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Attending anesthesiologist, National Taiwan University Hospital
Other Study IDs: 202504081RINA
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia; Swallowing Muscles
Keywords: dysphagia; noninvasive monitor; hypophayngeal muscles
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients without dysphagia: patients with dysphagia
- patients with dysphagia: patients with dysphagia

SUMMARY:
This project aims to develop a non-invasive monitoring approach using wearable devices, with validation against high-resolution impedance manometry. We plan to recruit 20 healthy participants aged 20-50 years and 20 patients with dysphagia. Patients will first undergo swallowing endoscopy to assess their swallowing status. Electromagnetic near-field coupling technology will then be applied to collect muscle contraction data during swallowing. A wearable sensor attached to the neck will provide detailed dynamic data on swallowing muscle activity to support clinical applications. Validation will be performed using high-resolution impedance manometry. In addition, anthropometric measurements, biochemical tests, and swallowing-related questionnaires will be collected. Statistical analysis will be used to examine correlations between measurement modalities and validate the effectiveness of the developed wearable technology.

DETAILED DESCRIPTION:
As Taiwan enters a super-aged society in 2025, the number of elderly patients with multiple comorbidities is rapidly increasing, and the risk of dysphagia rises with advancing age. Due to neuronal degeneration and muscle atrophy, elderly patients often experience slower recovery of swallowing ability after general anesthesia, sometimes requiring up to seven days to return to baseline function. Therefore, postoperative monitoring of swallowing function and timely rehabilitation interventions are essential to reduce complications and facilitate early discharge. Traditional swallowing assessment methods, such as videofluoroscopic swallowing study and high-resolution manometry, provide valuable information but are limited by radiation exposure and invasiveness. Hence, the development of non-invasive swallowing measurement devices is of great importance.

This project aims to develop a non-invasive monitoring approach using wearable devices, with validation against high-resolution impedance manometry. We plan to recruit 20 healthy participants aged 20-50 years and 20 patients with dysphagia. The patients will first undergo Videofluoroscopic Swallow Study (VFSS) or swallowing endoscopy to assess their swallowing status. Electromagnetic near-field coupling technology will then be applied to collect muscle contraction data during swallowing. A wearable sensor attached to the neck will not only capture heart rate and respiratory rate but also provide detailed dynamic data on swallowing muscle activity to support clinical applications. Validation will be performed using high-resolution impedance manometry. In addition, anthropometric measurements, biochemical tests, and swallowing-related questionnaires will be collected. Statistical analysis will be used to examine correlations between measurement modalities and validate the effectiveness of the developed wearable technology.

This study is expected to provide a breakthrough in swallowing function monitoring and contribute to improving postoperative recovery in elderly patients. Ultimately, it may offer novel strategies for managing dysphagia in an aging society.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteer groups: (I) Healthy participants aged over 20 years; (II) Body mass index (BMI) between 18.5 and 30.

Inclusion criteria for patients with dysphagia: Penetration-Aspiration Scale (PAS) score > 1 on fiberoptic endoscopic evaluation of swallowing (FEES), and a PAS score > 1 when swallowing two boluses of IDDSI level 0 (thin liquid) consistency. A total of 20 patients was planned for enrollment.

Exclusion Criteria:

* (I) Current use of any medication that affects gastrointestinal motility;
* (II) History of gastrointestinal surgery.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will have no symptoms of dysphagia, whereas patients with dysphagia will undergo fiberoptic endoscopic evaluation of swallowing, with a Penetration-Aspiration Scale (PAS) score greater than 1.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
hypopharyngeal mean peak pressure | 5 minutes
  hypopharyngeal muscle contraction

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to ethical issue